CLINICAL TRIAL: NCT00876304
Title: Phase 1, Investigator And Subject-Blind, Placebo-Controlled, Randomized, Sequential Group, Multiple Ascending Dose Study To Assess The Safety, Tolerability, Pharmacokinetics And Pharmacodynamics Of PF-04802540 In Patients With Schizophrenia
Brief Title: Multiple Dose Safety Study of PF-04802540 in Subjects With Schizophrenia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Taisho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Taisho Pharmaceutical Co., Ltd.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: B0911004
Record Dates: First submitted 2009-04-03; First posted 2009-04-06 (Estimated); Last update posted 2010-03-19 (Estimated); Status verified 2009-10

CONDITIONS: Schizophrenia
Keywords: PF-04802540 multiple dose safety study
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- PF-04802540 (Experimental)
  Interventions: Drug: PF-04802540
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-04802540 — Multiple ascending doses for 10 days; planned doses include capsules totaling 5 mg and 20 mg every 12 hours, with additional doses determined based on accumulating data
  Arms: PF-04802540
Drug: Placebo — Placebo capsules every 12 hours for 10 days
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and pharmacokinetics of multiple ascending doses of PF-04802540 administered orally to subjects with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Males or females of non-childbearing capacity aged 18 to 55 years inclusive
* DSM-IV diagnosis of schizophrenia, stable symptoms for at least 3 months
* Body mass index in the range of 18 to 40 kg/m2 and body weight>45 kg.

Exclusion Criteria:

* Evidence or history of a primary DSM IV axis I diagnosis other than schizophrenia.
* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease
* Any condition possibly affecting drug absorption (eg, gastrectomy).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2009-04; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Safety assessments: vital signs, ECG, physical examination, laboratory tests, Columbia - Suicide Severity Rating Scale | 22 days
Adverse Events | 22 Days
Plasma concentrations of PF 04802540 and its metabolite, PF 04831035 | 12 Days

SECONDARY OUTCOMES:
Positive and Negative Syndrome Scale | 16 days
Clinical Global Impression of Severity and Improvement | 16 days
Extrapyramidal Symptom Rating Scale - Abbreviated | 16 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Glendale, California, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B0911004&StudyName=Multiple%20Dose%20Safety%20Study%20of%20PF-04802540%20in%20Subjects%20With%20Schizophrenia